CLINICAL TRIAL: NCT04445922
Title: Bioequivalence of Oral Formulations of Anastrozole in Healthy Chinese Volunteers Under Fed Condition: A Open-label, Randomized,Single- Dose,Two-period, Two-group, Crossover Study
Brief Title: Bioequivalence of Oral Formulations of Anastrozole in Healthy Chinese Volunteers Under Fed Condition
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TG1915ANA
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test-anastrozole tablet (Experimental): 1 mg anastrozole was produced and provided by Salutas Pharma GmbH
  Interventions: Drug: test-anastrozole tablet (Salutas Pharma GmbH)
- reference-anastrozole tablet (Experimental): 1 mg anastrozole was produced by AstraZeneca Pharmaceuticals LP.
  Interventions: Drug: reference-anastrozole tablet

INTERVENTIONS:
Drug: test-anastrozole tablet (Salutas Pharma GmbH) — Subjects were allocated to one of two groups randomly and equally with a 21-day washout interval between the two periods.All of them were randomized (1:1) to receive anastrozole as a single oral dose of the test drug or a single 1.0-mg oral dose of Arimidex
  Arms: test-anastrozole tablet
Drug: reference-anastrozole tablet — Subjects were allocated to one of two groups randomly and equally with a 21-day washout interval between the two periods.All of them were randomized (1:1) to receive anastrozole as a single oral dose of the test drug or a single 1.0-mg oral dose of Arimidex
  Other Names: Arimidex
  Arms: reference-anastrozole tablet

SUMMARY:
An open-label, randomized, two-period, two-group, crossover study was conducted in 26 healthy Chinese volunteers under fed conditions to assess the bioequivalence between two formulations of Anastrozole.

DETAILED DESCRIPTION:
Anastrozole is currently used as first-line treatment in locally advanced or metastatic breast cancer. A generic anastrozole tablet was developed to offer an alternative to the marketed tablet formulation.The aim of the current study was to evaluate the bioequivalence between the test and reference formulations of anastrozole in a single-dose, 2-period, 2-sequence crossover study with a 21-day washout interval. A total of 26 healthy Chinese female subjects were randomized to receive a single dose of 1.0-mg test and reference formulations of anastrozole within 30 min after beginning the consumption of a recommended high-fat, high-calorie breakfast (150 calories from protein, 250 calories from carbohydrate, and 500-600 calories from fat; total calories approximately 800-1000).This was repeated two times, separated by a 21-day washout period.Blood samples (3 mL) for pharmacokinetic analysis were collected predose and 20min, 40min, 1, 1.5, 2, 2h20min, 2h40min, 3, 3.5, 4, 4.5, 5, 7, 12, 24, 48 and 72 hours postdose and were determined by a fully validated high-pressure liquid chromatography-tandem mass spectrometry method. The evaluated pharmacokinetic parameters, including Cmax, AUC0-t, AUC0-∞,were assessed for bioequivalence based on current guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Postmenopausal volunteers aged between 18 and 65 years old.
* The body mass index is in the range of 19.0-28.0 kg/m2 (including the critical value). The weight is not less than 45 kg.
* The subjects have no family planning within 6 months and could select contraceptive method.
* Subjects who had not any medical history of cardiovascular, digestive, respiratory, nervous, haemal diseases or hepatic/renal impairment.

Exclusion Criteria:

* Meet the diagnostic criteria for osteoporosis.
* Subjects with vaginal bleeding.
* blood donation, massive blood loss (#400mL) or enrolled in other clinical trials 3 months prior to screening.
* any use of other prescription drugs (including contraceptive) 28 days prior to medication for this study.
* any history of alcohol abuse in the recent 2 years or moderate drinkers (drink more 2 units per day or 14 units per week);
* smoking more than 5 cigarettes per day during the 3 months prior to screening;

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2020-07-04 (Estimated); Primary Completion 2020-08-03 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
the ratios of geometrical mean | 60 days
  The two preparations were considered bioequivalent if the 90% CIs of the ratios of the primary pharmacokinetics parameters were within the predefined acceptance range of 80%-125%.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Cao, doctor, Principal Investigator — the study director of phase I clinical research center
Locations (1):
- Phase I Clinical Research Center, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No